CLINICAL TRIAL: NCT01795560
Title: US Follow-up After Appendicitis Attack.
Brief Title: Follow up by US Following Hospitalization With Periappendicular Abscess Refusing to be Operated on Within a Few Weeks.
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Ahud Sternberg, MD, Hillel Yaffe Medical Center
Other Study IDs: 5-13
Record Dates: First submitted 2013-02-18; First posted 2013-02-20 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Disorder of Appendix
Keywords: Periappendicular abscess; Ultrasound

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Follow up via ultrasonic abdoman after patients who were giagnosed and treated as periappendicular abcess and refused to be operated later on in the "interval period ". To ass what occured to their appendics ?

DETAILED DESCRIPTION:
During the last 10 years patients were hospitalized and treated with antibiotics due to the diagnosis of periappendicular abcess. they were invited to be operate after wards -appendectomy, electively few weeks later on. All these patients refused to be operated. What happend to their appendics few months or years later on via ultrasonic abdomen view??

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed in the last 10 years suffering from periappendicular abcess.

Exclusion Criteria:

* after appendectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed in the last 10 years suffering from periappendicular abcess.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Size and Condition of the Appendix. | 6 months to 12 years following Appendicitis

CONTACTS AND LOCATIONS:
Overall Officials: Gershon Keren, MD, Principal Investigator — Hillel Yaffe Medical Center, Infectious Diseases Unit